CLINICAL TRIAL: NCT00155259
Title: Docetaxel by 1 Hour Infusion Followed by 24 Hour Infusion of Cisplatin Plus Capecitabine as Neoadjuvant Chemotherapy for Locally Advanced Breast Cancer
Brief Title: Docetaxel, Cisplatin and Capecitabine as Neoadjuvant Chemotherapy for Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 930607
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2005-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer , Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Docetaxel , Cisplatin , Capecitabine

INTERVENTIONS:
Drug: Docetaxel , Cisplatin , Capecitabine

SUMMARY:
The primary endpoint of this phase II trial is the objective response rate of the regimen. The secondary endpoints include treatment-related toxicity, progression free survival and overall survival and breast conserving rate.

DETAILED DESCRIPTION:
This is an open-label phase II trial designed to test the effect and toxicity profile of combination of docetaxel, cisplatin, and capecitabine in locally advanced breast cancer patients.Breast cancer is one of the leading causes of cancer death for women in Taiwan. Despite the advance in multidisciplinary treatment, a significant number of patients eventually develop metastatic disease, especially those who present with locally advanced breast cancer (LABC). LABC remains an important and challenging problem in practice. In LABC, treatment strategies that include neoadjuvant chemotherapy have several potential advantages: early initiation of systemic therapy, in vivo assessment of response, and downstaging of primary tumor and regional lymphatic metastases, which makes breast-conserving surgery an option for many. The potential theoretical shortcomings include delay in local treatment, introduction of drug resistance, and unreliability of clinical staging. In practice, the advantages have exceeded the disadvantages. Clinical trial has demonstrated that docetaxel and capecitabine is highly effective in the treatment of metastatic breast cancer. On the other hand, our previous study has demonstrated that combination of taxane and cisplatin is highly effective in the treatment of locally advanced and metastatic breast cancer. We design a combination chemotherapy using docetaxel with cisplatin and capecitabine in the treatment of locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with histological proven LABC, without metastasis, and no prior therapy. LABC is defined as follows：

  1. Tumor more than 5 cm in diameter
  2. Tumor involvement of chest wall (ribs or intercostals or serratus anterior muscles) or skin (ipsilateral cutaneous edema, ulceration, or satellite nodules)
  3. Clinical evident inflammatory carcinoma
  4. Ipsilateral fixed axillary adenopathy
* Measurable disease by physical examination, breast sonography and other image study
* KPS≧ 70%
* Adequate bone marrow reserve, defined as white blood cell (WBC)≧ 3,500/ mm3, absolute neutrophil count (ANC)≧ 1,500/mm3, platelets ≧ 100,000/mm3
* Adequate liver and kidney function: total bilirubin ≦ 2.0 mg/dl, serum alanine transaminases (ALT) and aspartate transaminase (AST) ≦ 3 times upper normal limit, serum creatinine ≦ 1.5 mg/dl
* Patients must be ≦ 65 years old
* Signed informed consent

Exclusion Criteria:

* Patients who have received prior treatment (including hormonal therapy, chemotherapy, radiotherapy or biological therapy) for LABC. Concomitant use of above therapy will no be allowed.
* Pregnant or lactating woman
* Metastases disease other than regional lymph node metastases (supraclavicular lymph node metastases is not eligible)
* Prior serious cardiac conditions such as angina, myocardial infarction, cardiomyopathy, severe cardiovascular disease or cardiac arrhythmias
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Secondary malignancy in past five years before entry of the study (except in situ carcinoma of the cervix, or adequately treated basal cell carcinoma of the skin)
* Active infection (at the discretion of the investigator)
* Significant neurological (such as seizures) or psychiatric disorder

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this phase II trial is the objective response rate of the regimen. | 2005~2006

SECONDARY OUTCOMES:
The secondary endpoints include treatment-related toxicity, progression free survival and overall survival and breast conserving rate. | 2005~2006

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, M.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan